CLINICAL TRIAL: NCT01245712
Title: Assessing the Cosmesis and Toxicity of Partial Breast Irradiation Using Proton Beam Irradiation
Brief Title: Radiation Therapy in Treating Patients With Stage 0-II Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0818; NCI-2011-01102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2009-0818 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Adenocarcinoma; Ductal Breast Carcinoma In Situ; Invasive Breast Carcinoma; Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (APBI) (Experimental): Within 10 weeks of last breast cancer surgery, patients undergo APBI delivered with proton radiation BID for 5 days.
  Interventions: Radiation: Accelerated Partial Breast Irradiation; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Radiation: Accelerated Partial Breast Irradiation — Undergo APBI delivered with proton radiation
  Other Names: APBI
Radiation: Proton Beam Radiation Therapy — Undergo APBI delivered with proton radiation
  Other Names: PBRT; Proton Radiation Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the side effects and how well radiation therapy works in treating patients with stage 0-II breast cancer. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the cosmesis, acute toxicity and late toxicity in patients treated with accelerated partial breast irradiation delivered with proton radiation.

SECONDARY OBJECTIVES:

I. To evaluate the convenience of accelerated partial breast irradiation and quality of life during accelerated partial breast irradiation.

II. To estimate the in-breast tumor control rates in patients treated with accelerated partial breast irradiation delivered with proton radiation.

III. Compare dosimetry to alternate treatment modalities.

OUTLINE:

Within 10 weeks of last breast cancer surgery, patients undergo accelerated partial breast irradiation (APBI) delivered with proton radiation twice daily (BID) for 5 days.

After completion of study treatment, patients are followed up at 6 weeks, 6 months, 1 year, and 18 months, then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

Women who satisfy all of the following conditions are the only patients who will be eligible for this study.

1. The patient must consent to be in the study and must have signed an approved consent form conforming with federal and institutional guidelines.
2. Patients must be >/= 18 years old. (Adenocarcinoma of the breast is not seen in children)
3. English and non-English speaking patient
4. The patient must have stage 0, I, or II breast cancer. If stage II, the tumor size must be 3 cm or less.
5. On histological examination, the tumor must be DCIS or invasive adenocarcinoma of the breast.
6. Surgical treatment of the breast must have been lumpectomy. The margins of the resected specimen must be histologically free of tumor (DCIS and invasive).

   Re-excision of surgical margins is permitted.
7. Gross disease must be unifocal with pathologic (invasive and/or DCIS) tumor size 3 cm or less. (Patients with microscopic multifocality are eligible as long as total pathologic tumor size is 3 cm or less.)
8. Patients with invasive breast cancer are required to have axillary staging which can include sentinel node biopsy alone (if sentinel node is negative), sentinel node biopsy followed by axillary dissection or sampling with a minimum total of 6 axillary nodes (if sentinel node is positive), or axillary dissection alone (with a minimum of 6 axillary nodes). Axillary staging is not required for patients with DCIS.
9. The target lumpectomy cavity must be clearly delineated and the target lumpectomy cavity/whole breast reference volume must be < 30% based on the postoperative/pre-enrollment CT scan.
10. Patients are eligible if, based on the postoperative CT scan, PBI is judged to be technically deliverable.
11. Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to enrollment and are deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

Exclusion Criteria:

Women with one or more of the following conditions also are ineligible for this study.

1. Men are not eligible for this study.
2. Individuals that are considered to be cognitively impaired.
3. T2 (> 3.0 cm), T3, stage III, or stage IV breast cancer.
4. More than 3 histologically positive axillary nodes.
5. Axillary nodes with definite evidence of microscopic or macroscopic extracapsular extension.
6. Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes at time of enrollment unless there is histologic confirmation that these nodes are negative for tumor.
7. Suspicious microcalcifications, or densities (in the ipsilateral or contralateral breast as documented on mammogram or breast ultrasound) unless biopsied and found to be benign.
8. Non-epithelial breast malignancies such as sarcoma or lymphoma.
9. Proven multicentric carcinoma (invasive cancer or DCIS) in more than one quadrant or separated by 4 or more centimeters.
10. Paget's disease of the nipple.
11. Synchronous bilateral invasive or non-invasive breast cancer.
12. Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation. (If surgical margins are rendered free of disease by re-excision, the patient is eligible.)
13. Clear delineation of the extent of the target lumpectomy cavity not possible.
14. Treatment plan that includes regional nodal irradiation.
15. Prior radiation to the index breast
16. Documented diagnosis of collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
17. Pregnancy or lactation at enrollment.
18. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Cosmesis Score | 1 year
  Patient-reported cosmesis score on the Breast Cancer Treatment Outcomes Scale (BCTOS) at 1 year. Cosmesis scores range from 1 (excellent) to 4 (poor), and scores of 3 (fair) or more indicate adverse cosmetic outcomes.

SECONDARY OUTCOMES:
Rate of CTCAE Grade 3+ Confluent Moist Desquamation | Within 6 weeks of radiation therapy
  Rate of CTCAE grade 3+ confluent moist desquamation estimated within 6 weeks of radiation therapy with a 90% credible interval. If we observe CTCAE grade 3+ confluent moist desquamation in only 20 patients, then our 90% credible interval will be 7% to 13%.
Percent of Patients with Local Failure | 10 years
  Percent of patients with local failure at 10 years estimated with an exact 95% confidence interval. If there is 1 patient with local failure at 10 years, and researchers have follow-up on all patients at 10 years, then the upper limit of the exact 95% confidence interval will be 2.8%. If researchers don't have 10 years of follow-up on all patients researchers will use the product-limit estimator of Kaplan and Meier (1958) to estimate the local failure rate at 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Mitchell, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org